CLINICAL TRIAL: NCT05552040
Title: Adaptation and Effectiveness of START NOW in the Treatment of Opioid Addicted Individuals Enrolled in Outpatient Based Opioid Treatment
Brief Title: START NOW in the Treatment of Opioid Addicted Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Robert L Trestman, Professor and Chair, Department of Psychiatry and Behavioral Medicine, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-20-1064
Record Dates: First submitted 2022-09-14; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: START NOW group psychotherapy versus Treatment-as-Usual group psychotherapy in OUD individuals in an OBOT program
Who Masked: Outcomes Assessor
Masking Description: Statistical analysis completed by Virginia Tech Department of Statistics faculty and graduate students who were all blinded with respect to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- START NOW Group (Experimental): START NOW is an evidence-informed psychotherapy composed of a total of 32-skills-based-sessions, originally designed for inmates in correctional systems. A previous study of incarcerated individuals found that for each additional session of START NOW completed, a 5% reduction in the incident rate of disciplinary reports was noted.10 In fact, individuals with a higher overall security risk score also had a greater reduction in the number of disciplinary reports with more sessions attended, suggesting that START NOW is an effective behavioral intervention for those who need it most. A follow-up study on these same participants concluded that START NOW appears to have a beneficial clinical effect with each session completed being associated with a 5% decrease in subsequent psychiatric hospital days.
  Interventions: Behavioral: START NOW Group
- Treatment-as-Usual (TAU) Group (Active Comparator): TAU groups are weekly sessions required in an OBOT clinic and focus primarily on supportive therapeutic techniques.
  Interventions: Behavioral: START NOW Group

INTERVENTIONS:
Behavioral: START NOW Group — START NOW psychotherapy is a CBT, DBT and skills-based intervention

SUMMARY:
This investigation involves a partially randomized clinical trial examining the effectiveness of combining buprenorphine/naloxone MAT with START NOW, a skills-based psychosocial intervention modified specifically for the ambulatory substance use disorder (SUD) patient population. START NOW is an integrated evidence-informed model based on an adapted form of dialectical behavior therapy (DBT), a type of cognitive behavior therapy (CBT) with promising indications for treating SUD as it targets impulsive and self-destructive behaviors. Furthermore, START NOW combines CBT, the most widely used evidence-based psychosocial intervention for treating mental disorders, with motivational interviewing, which in clinical trials has been shown to be an effective technique for engaging patients with SUD. In addition to tracking clinical outcomes such as abstinence rates through weekly urine drug screens, this investigation will use: clinician assessments of disease severity, researcher-evaluated tests of delayed discounting (DD) and demand tasks, and self-report surveys assessing impulsivity, aggression, interpersonal skills, and other measures to capture the patients' sense of progress in treatment in regards to their substance use, health, lifestyle, and community. By using DD and functional magnetic resonance imaging (fMRI), the identification of the neural correlates of START NOW treatment response will begin to elucidate the mechanisms of START NOW's effects and more. This investigation's outcome measures may not only compare the effectiveness between START NOW and treatment-as-usual (TAU), but also provide a more realistic, holistic view of patients and their well-being throughout the recovery process.

DD will be performed by both START NOW group members and TAU group members at their group therapy meetings as per protocol. Additionally, START NOW group members randomized and consented to have an fMRI will also perform DD before the scan is initiated.

DETAILED DESCRIPTION:
There is an unmet need for implementing a clinically superior behavioral therapy intervention for medication-assisted treatment of opioid use disorder.

One strategy for fighting the opioid epidemic is to improve treatment and detoxification programs. In the United States, the Drug Addiction Treatment Act of 2000 requires that physicians combine medication-assisted treatment (MAT) with a behavioral intervention. However, there is no clear evidence regarding what form of therapy is most effective when coupled with MAT for opioid use disorder (OUD) management.

This investigation will explore the impact of a novel skills-based psychosocial intervention called START NOW, which has been modified for the substance use disorder (SUD) patient population. The promising therapeutic potential of START NOW is evident in the growing data affirming the program's utility and the psychosocial techniques with substantial supportive evidence incorporated into the program. This investigation will attempt to prove through a number of clinical and behavioral parameters how START NOW with MAT may be an effective treatment program for patients undergoing OUD treatment.

START NOW is an evidence-informed psychotherapy composed of a total of 32-skills-based-sessions, originally designed for inmates in correctional systems. A previous study of incarcerated individuals found that for each additional session of START NOW completed, a 5% reduction in the incident rate of disciplinary reports was noted. In fact, individuals with a higher overall security risk score also had a greater reduction in the number of disciplinary reports with more sessions attended, suggesting that START NOW is an effective behavioral intervention for those who need it most. A follow-up study on these same participants concluded that START NOW appears to have a beneficial clinical effect with each session completed being associated with a 5% decrease in subsequent psychiatric hospital days. Evidence continues to build in support for START NOW as a behavioral intervention as its implementation continues to grow. For example, START NOW is currently being used in correctional facilities in more than 10 states in the US. Using a randomized, controlled trial in Europe, investigators are evaluating START NOW's ability to enhance psychosocial adjustment and well-being and to reduce oppositional and aggressive behavior in 128 institutionalized female adolescents diagnosed with oppositional defiant disorder and/or conduct disorder.

Investigators hypothesize that OUD patients who complete START NOW group therapy will show a statistically greater reduction in impulsivity, delay discounting, and illicit drug use compared to the OUD patients who complete the treatment-as-usual (TAU) because of START NOW's integrated model of care. For example, START NOW combines CBT, the most widely used evidence-based psychosocial intervention for treating mental disorders, with motivational interviewing, which in clinical trials has been shown to be an effective conjunction intervention for SUD. START NOW exercises psychosocial techniques similar to dialectical behavior therapy (DBT), a type of cognitive behavior therapy (CBT) with promising indications for treating SUD because it targets impulsive and self-destructive behaviors. A currently unpublished pilot study using START NOW in an office-based outpatient treatment setting with OUD yielded patient satisfaction data and detailed feedback; this data is being used to guide the modification process of START NOW's materials and delivery so that START NOW is more culturally sensitive and appropriate for the SUD patient population. This proposed investigation will use the revised START NOW participant workbooks and real-life exercises adapted specifically for SUD.

Investigators believe that START NOW possesses many components that make it a particularly useful behavioral intervention for SUD. For example, the program is divided into four units, and Unit 1, while teaching focusing skills and functional analysis of behavior skills, tries to teach individuals how to develop self-control, cope with stressors, and become ready for change. Unit 2 focuses on understanding and coping with feelings and emotions. Unit 3 aims to teach individuals how to build positive relationships with others. Finally, Unit 4 focuses on setting and reaching personal goals. Investigators hypothesize that using START NOW's manual-guided approach will confer improved executive functioning skills and decreased delayed discounting, which will ultimately yield better clinical outcomes. This will be the first investigation evaluating an adapted START NOW for treating OUD with buprenorphine/naloxone MAT in the outpatient setting. The study aims to provide clinical utility for healthcare professionals in the field of addiction medicine and contributions to the understanding of addiction biology.

Delayed discounting may be a useful biomarker for tracking and predicting clinical outcomes for patients undergoing rehabilitation Delayed discounting (DD) is a behavioral marker for impulsive decision-making and devaluation of delayed rewards. This investigation will use delayed discounting as an objective measure of cognitive executive functioning of its study participants before, during, and after treatment. Furthermore, we will compare DD values to clinical outcomes, clinician assessments, and self-report assessments in order to see if there is a correlation between all of these measures.

Opiate addiction has consistently been found to correlate with delay discounting, especially during periods of active addiction and especially amongst intravenous heroin users. However, methadone treatment, even when it resulted in the avoidance of relapse or other drug use, did not significantly improve delay discounting, when compared to the treatment condition in which participants continued to abuse substances. The authors of this study suggest that this may be due to patients receiving effective drug treatment that does not involve prolonged substitution therapy may be forced to develop better self-control skills to remain abstinent. In a comparison between buprenorphine and methadone, a 2012 study found buprenorphine has a number of advantages over methadone for use in MAT. While methadone is a full agonist of opioid receptors, buprenorphine is a weak partial agonist, especially at the mμ opioid receptor, thereby causing less analgesia and euphoria.

Investigators hypothesize that methadone, as a full agonist more prone to inducing euphoria and thereby enabling drug abuse, may prevent the improvement in cognitive executive functions theorized to be impaired by substance dependence. Moreover, the unique pharmacokinetics and pharmacodynamics profiles of buprenorphine may allow for more stable disease control, reduced harmful behavior, and thus improvements in cognitive executive functions (namely DD) for individuals undergoing concomitant buprenorphine MAT and an effective psychosocial intervention such as START NOW. Furthermore, previous studies found that DD decreases in individuals completing treatment for opioid dependence with buprenorphine MAT, but they failed to find any relationship between DD measures and abstinence outcomes.

While DD might be a stable trait in some individuals, a technology of behavior that manipulates DD may not only impact DD but also reduce the impulsive choices that comprise behavioral patterns of addiction and poor health-decision-making. Studies have successfully shown reduced delay discounting (DD) when targeting cognitive skills such as learning to activate one's working memory for longer periods. The clinical trial proposed by this investigation not only utilizes MAT and START NOW as a unique approach for not only treating OUD and developing effective clinical practices, but also aims to enhance the understanding of DD in addiction treatment outcomes. Showing a correlation between DD and opioid addiction may enable clinicians and researchers alike with the ability to predict treatment success and to use DD as a biomarker for OUD disease regression or relapse.

DD will be measured in both groups during the appointed time at the designated group sessions. Those in the START NOW group that have been randomized to have the fMRI will also perform DD before their fMRI scan.

Neural correlates will be studied from before and after the START NOW treatment begins. Neural correlates in the TAU group will be not studied. The identification of the neural correlates of START NOW treatment response may lead to a number of potential future directions. First, understanding who is most likely to respond to treatment may help target treatment efforts. Second, this information will help elucidate the mechanisms of START NOW effects, allowing for refining and further development of the treatment approach. Third, future efforts could use knowledge gained in this proposal to directly target behavior change with techniques such as transcranial magnetic stimulation or real-time fMRI biofeedback. All of the information obtained through this investigation's outcome measures may help in the development of a superior behavioral intervention for OUD and improve our understanding of addiction biology.

For participants in the START NOW group, those that are eligible and interested will be randomized to have an fMRI or not. Only 20 participants will complete the fMRI. These participants will perform delayed discounting tasks in fMRI sessions before and after behavioral intervention. Investigators expect the neural correlates of delayed discounting to predict START NOW treatment success. Depending on the results, the fMRI component of this investigation may elucidate the mechanisms of START NOW's effects, help create a model for predicting treatment success, or provide information on how to better target behavior change. Neural correlates will only be studied in the START NOW group, comparing before and after the treatment begins.

Beyond capturing a participant's drug use and clinical disease course, this study aims to capture participants' personal satisfaction with one's livelihood and other measures to effectively compare START NOW with TAU. Moreover, investigators hypothesize that in the best-case scenario, individuals who maintain their sobriety, regardless of the behavioral treatment intervention they receive, will show improvements in other aspects of their lives. For example, individuals who remain sober throughout treatment (clean urine drug screens) will also show: decrease disease severity (CGI-S), increased disease improvement (CGI-I), reduced impulsivity (BIS), decreased aggression (AGQ), and fewer interpersonal problems (IIP). With all of these measures, investigators hope to offer a more compassionate, comprehensive view-one that extends beyond the disease and diagnosis-of the whole patient.

Data Analysis For Specific Aim 1, the differences between START NOW and TAU utilizing an intent-to-treat model with a regression statistical approach will be evaluated. The specific regression model will be determined by the distribution of the data. For Specific Aim 2 and 3, self-assessment by the participants between START NOW and TAU will be compared in the stated domains using an analysis of variance model (ANOVA). For Specific Aim 4, neural correlates associated with delay discounting task performance will be compared between groups. For Specific Aim 5, variance / co-variance matrixes of SNAP compared to the BIS, AGQ, and IPP will be looked at to determine the factor structure and correlation between the instruments.

Investigators hypothesize that activation of valuation networks (e.g., dopaminergic networks connecting midbrain to frontal cortices) will predict and change in response to START NOW treatment success.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older with OUD diagnosis participating in OBOT

Exclusion Criteria:

1. Imminent suicide risk at investigator discretion
2. Unable to commit to participation in the planned 32 session regimen
3. Unmanaged psychiatric illness that would interfere in study participation, as determined by investigator
4. Pregnant patients with OUD [for the imaging study ONLY]

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Retention in treatment by group attendance | 32 -52 weeks
  Translates to # groups attended (max 32)
Retention in treatment by time in study | 32 -52 weeks
  Weeks from consent to last group attended
Intensity of treatment | 32 -52 weeks
  total number-of-groups-attended divided by number of weeks from consent to last group attended
Drug use based on drug screen results | 32-52 weeks
  Drug use during trial period was determined by drug screens, which were collected weekly or monthly based on clinician preference throughout the entire 8-month investigation for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Trestman, PhD, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No